CLINICAL TRIAL: NCT00500097
Title: Diabetic Retinopathy and Diabetic Macular Edema Screening by Non-Physicians With Limited Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Thailand (Other Government)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 0321/1874
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ophthalmoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Digital retina image
Device: direct ophthalmoscopy
Procedure: comprehensive eye exam

SUMMARY:
The purpose is to assess accuracy of digital retinal image interpretation by technicians and direct ophthalmoscopy by nurses for the determination of diabetic retinopathy severity and the presence of diabetic macular edema for the identification of referrals to ophthalmologists. The results of both screening methods were compared with comprehensive eye examination by ophthalmologists.

DETAILED DESCRIPTION:
Diabetic visual disabilities have increasingly become a global concern since a number of diabetic patients are expected to surge dramatically in the coming decade. Essential means to minimize this problem are detecting vision-threatening diabetic retinopathy early in the course of disease and timely interventions by ophthalmologists.

The American Diabetes Association had issued a guideline for the detection and recommended regular comprehensive eye examination as a preferred method. However, it is not likely that there will be ophthalmologists enough to comprehensively examine the surging number of diabetic patients. Other practical screening methods, such as an interpretation of digital retinal images or direct ophthalmoscopy employed by other health care providers, for identifying the retinopathy for referral to ophthalmologists, should minimize this problem.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients defined by WHO criteria
* lived in the geographic area of participated hospitals

Exclusion Criteria:

* have contraindications for receiving mydriatic medications
* have ocular media not clear enough for making diagnosis by any of the screening equipment
* have other retina diseases precluded the diagnosis of diabetic retinopathy

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2005-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, kappa coefficient | cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Paisan Ruamviboonsuk, MD, Principal Investigator — Department of Ophthalmology, Rajavithi Hospital, Bangkok, Thailand 10400
Locations (1):
- Department of Ophthalmology, Rajavithi Hospital, Bangkok, Thailand